CLINICAL TRIAL: NCT05070091
Title: The Impact of Pituitary-thyroid and Pituitary-adrenal Axes Function on COVID-19 Clinical Course.
Acronym: ENDO-COVID19
Status: Completed | Type: Observational
Sponsor: Medical University of Gdansk (Other)
Collaborators: National Center for Research and Development, Poland (Other)
Responsible Party: Sponsor
Other Study IDs: ENDO-COVID19
Record Dates: First submitted 2021-10-04; First posted 2021-10-06 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: COVID-19; Low Triiodothyronine Syndrome; Adrenal Insufficiency; Subacute Thyroiditis; Hypothyroidism; Hyperthyroidism
Keywords: COVID-19, thyroid, adrenal gland, pituitary, glucocorticoids
MeSH Terms: conditions — COVID-19; Euthyroid Sick Syndromes; Adrenal Insufficiency; Thyroiditis, Subacute; Hypothyroidism; Hyperthyroidism; Thyroid Diseases; Pituitary Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main focus of the study is the assessment of hormonal function in the course of COVID-19 infection with special regard for trends predicting clinical events defined as primary endpoints of the study.

ELIGIBILITY:
Inclusion Criteria:

* PCR-confirmed COVID-19 infection
* volunteers consenting to participate

Exclusion Criteria:

* no consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with PCR-confirmed COVID-19 infection.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Meeting the primary endpoint criteria. | Time of hospitalization, typically less than one month.
  Primary endpoint is defined as a composite endpoint including death, mechanical ventilation, vasopressor use, noninvasive ventilation, prolonged hospital stay (>10 days).

CONTACTS AND LOCATIONS:
Overall Officials: Renata Świątkowska-Stodulska, MD PhD, Study Director — Medical University of Gdansk; Agata Berlińska, MD, Principal Investigator — Medical University of Gdansk
Locations (2):
- Poland (2):
  - 7 Szpital Marynarki Wojennej, Gdansk
  - Medical University of Gdansk, Gdansk